CLINICAL TRIAL: NCT06810284
Title: Effect of Sildenafil in Association to Hypothermia on Survival Without Brain Lesions in Term Neonates with Hypoxic-ischemic Encephalopathy (SHINE): Pharmacokinetic Study - Step 1
Brief Title: Sildenafil Plus Hypothermia to Treat Neonatal Encephalopathy
Acronym: SHINE1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P180603; 2023-508928-35-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-24; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-01

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: Hypoxic-ischemic encephalopathy; Sildenafil; Neuroprotection; newborn
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- intervention group (Experimental): Controlled hypothermia + open-label IV Sildenafil
  Interventions: Drug: Sildenafil Citrate (IV)

INTERVENTIONS:
Drug: Sildenafil Citrate (IV) — Controlled hypothermia initiated before 6h after birth (servo-controlled 33.5°C during 72h followed by a 12-h rewarming period up to 36.5°C), open-label IV Sildenafil Citrate (Revatio®, 10 mg/12.5 mL, Pfizer) 0.4 mg/kg delivered over 3 hours, followed by a maintenance infusion at 1.6 mg/kg/day for 72h
  Other Names: Revatio

SUMMARY:
The main objective of this study is to assess pharmacokinetics features of IV sildenafil in neonates with hypoxic-ischemic encephalopathy and treated by controlled hypothermia. This phase 2 study will prepare a large phase 3 randomized controlled trial to demonstrate the superiority of a combinatory therapy associating IV sildenafil and controlled hypothermia compared to Placebo and controlled hypothermia, on survival without brain lesions on MRI at discharge, in neonates born after 36 weeks of gestation.

DETAILED DESCRIPTION:
Neonatal hypoxic-ischemic encephalopathy (HIE) following birth asphyxia is a major cause of death or long-term disability in term neonates, affecting about 1-4 per 1.000 live births and consequently 30.000 infants/year in Europe. Incidence and consequences of HIE are even more common and severe in less privileged settings, affecting about 1 million infants every year worldwide.

In recent years, therapeutic hypothermia became the standard of care to improve outcomes after perinatal hypoxic-ischemic insults. Despite hypothermia and state-of-the-art neonatal intensive care, 45-50% of children with moderate or severe HIE (i.e., 12.000 - 15.000 infants/year in Europe) still die or suffer from long-term neurodevelopmental impairment. Therefore, additional early neuroprotective interventions, beside hypothermia, are warranted to further improve the outcomes of HIE.

The best conceivable treatment for HIE is the restoration of cerebral blood flow (CBF) as soon as possible because its decrease 12-24 hours indicates poor prognosis in term newborns with HIE in human and rodents. Recently, the inhalation of nitric oxide (NO) has been found to be beneficial in several preclinical models of ischemia, but NO-dosage and time period of exposure seem to be crucial for beneficial effects. Another option that enhances the effects of endogenous NO is to increase the cyclic guanosine monophosphate (cGMP) concentration by blocking its degradation by phosphodiesterases (PDEs). In particular, sildenafil, a potent selective PDE-5 inhibitors, prolong the action of cGMP in multiple vascular territories. Recent findings strongly indicate that sildenafil citrate treatment induced a significant increase in CBF, reduces HI damage and improves motor locomotion in neonatal rats. In addition, anti-inflammatory effects of sildenafil may provide protection against lesion extension in the late phase after brain ischemia in neonatal mice. Together, these data strongly suggest that sildenafil, already used in neonatal pulmonary hypertension - a co-morbid condition that could worsen brain injury - may represent an interesting therapeutic strategy for neonatal neuroprotection. SHINE project aims to test its added value in addition to hypothermia to prevent neonatal death and brain damage following HIE. Pharmacokinetics (PK) data from oral administration suggest that serum concentrations within therapeutic targets are achieved with a dosage corresponding to the bioavailability of oral sildenafil under therapeutic hypothermia. However, plasma concentrations of continuous IV sildenafil infusion in neonates under hypothermic conditions with HIE has never been analysed justifying a PK study. This PK study sildenafil is mandatory to (i) ensure that the a priori IV dose determined as biologically effective remains within the therapeutic target with metabolic et PK changes potentially induced by both HIE condition and controlled hypothermia, (ii) ensure the absence of overdose and/or side effects of this dosage, at any time of the hypothermia treatment and rewarming, and (iii) adjust, if necessary, the dosage to reach the therapeutic target.

The investigators will perform a phase 2 pharmacokinetics observational study of IV sildenafil in neonates with HIE and exposed to controlled hypothermia (33.5°C) to ensure the safety and confirm the relevance of the sildenafil IV dose to be given in infants with hypothermia in the Phase 3 trial.

The pharmaco-statistical analysis will be conducted using non-linear mixed effects modeling to calculate the PK parameters of sildenafil as well as the inter-individual and the residual variabilities.

ELIGIBILITY:
Inclusion Criteria:

* 1/Neonates born at or after 36 weeks' gestation, treated by therapeutic servo-controlled hypothermia for neonatal hypoxic ischemic encephalopathy.

Therapeutic hypothermia should be decided according to French national guidelines.

* 2/ Social security coverage
* 3/ Informed consent of one of the two holders of parental authority.

Exclusion Criteria:

* 1/ Chromosomal aberrations and major malformations evidenced after birth
* 2/ Decision for "comfort care only" before study drug administration,
* 3/ Uncontrolled hemorrhagic syndrome,
* 4/ Severe hemodynamic failure at initiation, requiring at least two therapies (including either volume expansion, hydrocortisone or inotropes)
* 5/ Known hypersensitivity to the active substance or to any of the excipients
* 6/ Concomitant administration of nitrates or nitric oxide donors, Inhaled Nitric Oxide, other PDE5 inhibitors, inhibitors of CYP3A4
* 7/ Participation in another interventional study

Max Age: 12 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Plasma concentrations of Sildenafil within the first 5 days following treatment initiation. | From 3 hours after initiation of sildenafil and 48 hours after end of maintenance continuous infusion
  Pharmacokinetics features of IV sildenafil in neonates with HIE and treated by controlled hypothermia.

SECONDARY OUTCOMES:
Estimated clearance parameters | From initiation of sildenafil and 48 hours after end of maintenance continuous infusion
  Pharmacokinetics features of IV sildenafil in neonates with HIE and treated by controlled hypothermia.
volumes of distribution for IV sildenafil (l) | From initiation of sildenafil and 48 hours after end of maintenance continuous infusion
  Pharmacokinetics features of IV sildenafil in neonates with HIE and treated by controlled hypothermia.
Area under the plasma sildenafil concentration-time curve | From initiation of sildenafil and 48 hours after end of maintenance continuous infusion
  Pharmacokinetics features of IV sildenafil in neonates with HIE and treated by controlled hypothermia.
Maximum plasma sildenafil concentration achieved (individual exposure) | From initiation of sildenafil and 48 hours after end of maintenance continuous infusion
  Pharmacokinetics features of IV sildenafil in neonates with HIE and treated by controlled hypothermia.
Brain damage-free survival at hospital discharge on MRIs performed between 3.5 to 5 days and/or 10-30 days | between 3.5 to 5 postnatal days
  Brain damage-free survival at hospital discharge on MRIs performed between 3.5 to 5 days and/or 10-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BAUD, MD, PhD, Study Director — Hôpitaux Universitaires de Genève et Inserm U1141, Paris
Locations (1):
- Unité de Recherche Clinique, Entrepôts de données et Pharmacologie GHU Paris Centre, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yazdani A, Howidi B, Shi MZ, Tugarinov N, Khoja Z, Wintermark P. Sildenafil improves hippocampal brain injuries and restores neuronal development after neonatal hypoxia-ischemia in male rat pups. Sci Rep. 2021 Nov 11;11(1):22046. doi: 10.1038/s41598-021-01097-6. PMID 34764335
- [Background] Yazdani A, Khoja Z, Johnstone A, Dale L, Rampakakis E, Wintermark P. Sildenafil Improves Brain Injury Recovery following Term Neonatal Hypoxia-Ischemia in Male Rat Pups. Dev Neurosci. 2016;38(4):251-263. doi: 10.1159/000448327. Epub 2016 Sep 10. PMID 27614933
- [Background] Moretti R, Leger PL, Besson VC, Csaba Z, Pansiot J, Di Criscio L, Gentili A, Titomanlio L, Bonnin P, Baud O, Charriaut-Marlangue C. Sildenafil, a cyclic GMP phosphodiesterase inhibitor, induces microglial modulation after focal ischemia in the neonatal mouse brain. J Neuroinflammation. 2016 Apr 28;13(1):95. doi: 10.1186/s12974-016-0560-4. PMID 27126393
- [Background] Charriaut-Marlangue C, Nguyen T, Bonnin P, Duy AP, Leger PL, Csaba Z, Pansiot J, Bourgeois T, Renolleau S, Baud O. Sildenafil mediates blood-flow redistribution and neuroprotection after neonatal hypoxia-ischemia. Stroke. 2014 Mar;45(3):850-6. doi: 10.1161/STROKEAHA.113.003606. Epub 2014 Jan 28. PMID 24473179